CLINICAL TRIAL: NCT04515602
Title: Stratified Evaluation and Prediction of Survival Benefit for PDS or NACT-IDS in Advanced Ovarian Cancer, A Randomized, Phase 3 Trial After the SUNNY Study
Brief Title: Stratified Evaluation of PDS and NACT-IDS in Ovarian Cancer (FOCUS)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOCUS; SOC-4 (Registry Identifier: Shanghai Gynecologic Oncology Group); SGOG-OV6 (Registry Identifier: Shanghai Gynecologic Oncology Group)
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 Arm I (low/medium tumor burden) (Experimental): Primary debulking surgery with a maximal cytoreduction of complete gross resection within 3 weeks after biopsy, followed by at least 6 cycles of adjuvant chemotherapy and maintenance therapy for patients with gBRCA/sBRCA mutation, CR/PR after platinum-based therapy.
  Interventions: Procedure: Primary debulking surgery; Drug: PARPi
- Part 1 Arm II (low/medium tumor burden) (Active Comparator): Neoadjuvant chemotherapy with 3 cycles of chemotherapy, then followed by interval debulking surgery. The maximal time interval between course 3 chemotherapy and IDS is 6 weeks. And then 3 cycles of adjuvant chemotherapy and maintenance therapy for patients with gBRCA/sBRCA mutation, CR/PR after platinum-based therapy.
  Interventions: Procedure: Neoadjuvant chemotherapy; Drug: PARPi
- Part 2 Arm I (high tumor burden) (Experimental): Primary debulking surgery with a maximal cytoreduction of complete gross resection within 3 weeks after biopsy, followed by at least 6 cycles of adjuvant chemotherapy and maintenance therapy for patients with gBRCA/sBRCA mutation, CR/PR after platinum-based therapy.
  Interventions: Procedure: Primary debulking surgery; Drug: PARPi
- Part 2 Arm II (high tumor burden) (Active Comparator): Neoadjuvant chemotherapy with 3 cycles of chemotherapy, then followed by interval debulking surgery. The maximal time interval between course 3 chemotherapy and IDS is 6 weeks. And then 3 cycles of adjuvant chemotherapy and maintenance therapy for patients with gBRCA/sBRCA mutation, CR/PR after platinum-based therapy.
  Interventions: Procedure: Neoadjuvant chemotherapy; Drug: PARPi

INTERVENTIONS:
Procedure: Primary debulking surgery — Primary debulking surgery with a maximum cytoreduction, then followed by 6 cycles of Paclitaxel 175mg/m2 or Docetaxel 60-75 mg/m2 plus Carboplatin AUC (area under the curve) 5.
  Other Names: PDS
  Arms: Part 1 Arm I (low/medium tumor burden); Part 2 Arm I (high tumor burden)
Procedure: Neoadjuvant chemotherapy — 3 cycles of Paclitaxel 175mg/m2 or Docetaxel 60-75 mg/m2 plus Carboplatin AUC (area under the curve) 5, Interval debulking surgery with a maximal cytoreduction of complete gross resection, then followed by another 3 cycles of chemotherapy.
  Other Names: Neoadjuvant chemotherapy followed by interval debulking surgery, NACT-IDS
  Arms: Part 1 Arm II (low/medium tumor burden); Part 2 Arm II (high tumor burden)
Drug: PARPi — For patients with gBRCA/sBRCA mutation and CR/PR after first-line chemotherapy, maintenance therapy of PARP inhibitors.

SUMMARY:
The purpose of this study is to answer the fundamental question 'The Optimal Timing of Surgery' in advanced ovarian cancer patients with different tumor burden, and to perform translational study.

DETAILED DESCRIPTION:
OBJECTIVES: Compare the efficacy and safety in patients with advanced ovarian cancer treated with NACT-IDS versus PDS, among different tumor burden groups. Compare survival benefit of PARPi therapy in patients treated with PDS or NACT-IDS.

OUTLINE: This is a randomized phase III multicenter study. Patients will receive upfront maximal cytoreductive surgery followed by at least 6 cycles of adjuvant chemotherapy or 3 cycles of neoadjuvant chemotherapy followed by interval debulking surgery, and then at least 3 cycles of adjuvant chemotherapy, and maintenance therapy of PARP inhibitor for patients with gBRCA/sBRCA mutation who had a complete or partial clinical response after platinum-based chemotherapy. Patients are followed every 3 months within the first 5 years, and then every 6 months.

PROJECTED ACCRUAL: A total of 410 patients will be accrued for this study within 3 years.

ELIGIBILITY:
For Part 1:

Inclusion Criteria:

1. Females aged ≥ 18 years.
2. Pathologic confirmed stage IIIC and IV epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma (diagnosis by biopsy or core needle biopsy*, laparoscopic biopsy is not recommended). * If core needle biopsy could not be performed, patients should satisfy the following conditions:

   1. the patient has a pelvic mass, and
   2. omental cake or other metastasis larger than 2 cm in the upper abdomen, or pathologic confirmed extra-abdominal metastasis (FIGO IV), and
   3. preoperative CA125/CEA ratio > 25. If CA125/CEA ratio ≤ 25, imaging or endoscopy is obligatory to exclude a primary gastric, colon, or breast carcinoma.
3. cPCI score ≤ 8.
4. Performance status (ECOG 0-2).
5. Good ASA score (1/2).
6. Adequate bone marrow, renal and hepatic function to receive chemotherapy and subsequent surgery:

   1. white blood cells >3,000/µL, absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL, hemoglobin ≥9 g/dL,
   2. serum creatinine <1.25 x upper normal limit (UNL) or creatinine clearance ≥60 mL/min according to Cockroft-Gault formula or to local lab measurement,
   3. serum bilirubin <1.25 x UNL, AST(SGOT) and ALT(SGPT) <2.5 x UNL.
7. Comply with the study protocol and follow-up.
8. Patients who have given their written informed consent.

Exclusion Criteria:

1. Non-epithelial ovarian malignancies and borderline tumors.
2. Low grade ovarian cancer.
3. Mucinous ovarian cancer.
4. cPCI score > 8.
5. Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ or breast carcinoma (without any signs of relapse or activity).
6. Any other concurrent medical conditions contraindicating surgery or chemotherapy that could compromise the adherence to the protocol.
7. Other conditions, such as religious, psychological and other factors, that could interfere with provision of informed consent, compliance to study procedures, or follow-up.

For Part 2:

Inclusion Criteria:

1. Females aged ≥ 18 years, and < 70 years.
2. Pathologic confirmed stage IIIC and IV epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma.
3. cPCI score ≥ 10.
4. For FIGO IVB patients, abdominal lesions should be confined to one lobe of liver parenchyma metastasis or splenic metastasis. All extra-abdominal metastases should be resectable, such as inguinal lymph nodes, solitary supraclavicular, retrocrural or paracardial nodes.
5. Good performance status (ECOG 0-1).
6. Good ASA score (1/2).
7. Adequate bone marrow, renal and hepatic function to receive chemotherapy and subsequent surgery.
8. Comply with the study protocol and follow-up.
9. Patients who have given their written informed consent.

Exclusion Criteria:

1. Non-epithelial ovarian malignancies and borderline tumors.
2. Low grade ovarian cancer.
3. Mucinous ovarian cancer.
4. Clear cell carcinoma.
5. cPCI score < 8.
6. Lung metastasis, diffused pleural metastasis, bone metastasis, metastasis of mediastinal lymph node, internal mammary node, or multiple extra-peritoneal lymph nodes.
7. Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ or breast carcinoma (without any signs of relapse or activity).
8. Any other concurrent medical conditions contraindicating surgery or chemotherapy that could compromise the adherence to the protocol.
9. Other conditions, such as religious, psychological and other factors, that could interfere with provision of informed consent, compliance to study procedures, or follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Participants will be followed for at least 5 years after randomization
  Time from randomization to the date of death from any cause or date of last contact

SECONDARY OUTCOMES:
Progression-free survival | Participants will be followed for at least 2 years after randomization
  Time from randomization to the date of first progressive disease or death, whichever occurs first or date of last contact
Post-operative complications | Participants will be followed up to 3 months after randomization
  The surgical complications will be evaluated at 30-day, 60-day, 90-day after upfront cytoreductive surgery or interval debulking surgery
Quality of life assessments | Participants will be followed for at least 12 months or death after randomization, whichever came first
  Quality of life (Qol) as measured by QOQ-C30
Quality of life assessments | Participants will be followed for at least 12 months or death after randomization, whichever came first
  Quality of life (Qol) as measured by FACT-O
Accumulating treatment-free survival | Participants will be followed for at least 5 years or death after randomization, whichever came first
  The overall survival time minus the total treatment time of surgery and chemotherapy after randomization, regardless of the targeted therapy
Time to first subsequent anticancer therapy | Participants will be followed for at least 2 years or death after randomization, whichever came first
  Time from the date of randomization to the starting date of the first subsequent anticancer therapy or death, whichever occurs first or date of last contact
Time to secondary subsequent anticancer therapy | Participants will be followed for at least 5 years or death after randomization, whichever came first
  Time from the date of randomization to the starting date of the second subsequent anticancer therapy or death, whichever occurs first or date of last contact
Progression-free survival 2 | Participants will be followed for at least 5 years or death after randomization, whichever came first
  Time from randomization to second progressive disease or death, which occurs first or date of last contact

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Obstetrics & Gynecology Hospital of Fundan University, Shanghai
  - Shanghai First Maternity and Infant Hospital, Shanghai
  - Shanghai Jiao Tong University School of Medicine Xinhua Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No